CLINICAL TRIAL: NCT04728555
Title: Evaluation of an Intervention by a Pedagogical Digital Game About Radiotherapy for Children With Cancer
Brief Title: Intervention of a Game About Radiotherapy for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Gunn Engvall, Ass. Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Children's RT Game 21-22
Record Dates: First submitted 2021-01-19; First posted 2021-01-28 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Anxiety State
Keywords: Children, cancer, psychosocial support, serious game
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: A non-blinded randomized waiting list control study
Masking Description: Non-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game before RT start (Experimental): Intervention of a digital game five days before start of RadioTherapy
  Interventions: Procedure: Game about radiotherapy
- Game after RT start (Experimental): Intervention of a digital game three days after start of RadioTherapy
  Interventions: Procedure: Game about radiotherapy

INTERVENTIONS:
Procedure: Game about radiotherapy — A digital pedagogical game about radiotherapy

SUMMARY:
Background: Radiotherapy (RT) can be stressful and challenging for children exposed to a highly technical environment with large radiation equipment and immobilization devices. A pedagogical digital game about RT has been developed. Children who have received RT participated in work-shops and contributed with their experiences and suggestions.

Aim: To explore whether the intervention with a pedagogical digital game facilitate understanding, choice of distraction, creation of a sense of calmness and self-efficacy prior to and during RT and to describe the children's and the parents experiences and use of the game as a pedagogical tool. Further, to investigate feasibility in terms of reach, usability and acceptability.

Method: A feasibility and prospective waiting list control design is planned by recruiting 60 children (5-14 years) and their parents, for randomization into two groups. The first group will receive the game five days before start of RT. All children will have standard information one day before RT. The second group will have access to the game three days after start of treatment. The effects of the game will be investigated before and during RT and between groups as they receive the game at different time. Children will answer questionnaires about self-assessed anxiety, understanding of the procedure, distraction strategies, self-efficacy to remain motionless. Statistical comparative and correlational analyses will be calculated. Interviews will be performed with 12 children and 24 parents. Changes and further development of the game will be implemented based on the results of the responses.

Significance: The game can support children to undergo RT and be used nationally to prepare for RT. Thus all children receive similar information regardless of where they live, and contribute to increased knowledge, autonomy, reduce fear and anxiety. In the long term, the use of anesthesia could decrease for children.

DETAILED DESCRIPTION:
Data Collection and procedure:

Access to the game for children randomized to the first group: Four to six days before start of treatment.

Questionnaires to all children: Questions about state and trait anxiety, and radiotherapy before the information meeting with the oncology nurse, one day before the start of treatment, at baseline.

Questionnaire to parents: Questions about state and trait anxiety before the information meeting with the oncology nurse at baseline.

Information meeting with all children and their parents: Information about radiotherapy by oncology nurse at baseline Questionnaires to all children: Questions about state anxiety and radiotherapy on treatment day one and three.

Access to the game for children randomized to the second group: Day three after start of treatment.

Questionnaire to all children: Questions about state anxiety on treatment day six and 15.

Questionnaire to all children: Questions about the digital game one week after access to the game.

Game logs: Collection of game logs one week after the intervention.

Interview of 12 children and 24 parents: Within four weeks after end of treatment.

Power: A power of 0.80, an alpha value of 0.05 and a size-effect of 0.5 provided an estimation of 26 participants in each group. Thirty participants are planned in case of dropouts.

Data analysis: Comparative and correlational statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

Children aged 5-14 years old who are going to have radiotherapy at the Skandion Clinic, Uppsala with or without sedation/anesthesia, understand and can speak Swedish and have access to a computer.

Exclusion Criteria:

Severe cognitive impairment and too seriously ill to be able to answer questions.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Children's State anxiety, change is being assessed | Baseline and on treatment day three, six and 15
  From the questionnaire STAI-C1

SECONDARY OUTCOMES:
Children's Trait anxiety | Baseline
  From the questionnaire STAI-C2
Children's self-efficacy to remain motionless, change is being assessed | Baseline and on treatment day three
  From a questionnaire made for the study
Children's perception of the digital game about radiotherapy: usability and engagement | One week after the intervention
  From the questionnaire PENS

OTHER OUTCOMES:
Parent's State and Trait anxiety | Baseline
  From the questionnaire STAI-Y1 and STAI-Y2

CONTACTS AND LOCATIONS:
Overall Officials: Gunn Engvall, Professor, Principal Investigator — Women's and Children's Health, Uppsala University, Sweden
Locations (1):
- Department of Women's and Children's Health, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Results will be reported in scientific journals

REFERENCES:
- [Background] Cederved C, Back J, Angstrom-Brannstrom C, Ljungman G, Engvall G. Co-creation of a Serious Game About Radiotherapy: Participatory Action Research Study With Children Treated for Cancer. JMIR Hum Factors. 2022 May 31;9(2):e34476. doi: 10.2196/34476. PMID 35639467
- [Background] Cederved C, Angstrom-Brannstrom C, Ljungman G, Engvall G. Parents' experiences of having their children take part in participatory action research creating a serious game about radiotherapy. Radiography (Lond). 2023 Jan;29(1):95-100. doi: 10.1016/j.radi.2022.10.005. Epub 2022 Oct 29. PMID 36327521